CLINICAL TRIAL: NCT01172977
Title: Neurological Complications at Stroke Patients With Diabetes Mellitus During the First Six Months After a Cerebral Ischemia
Brief Title: Neurological Complications at Stroke Patients With Diabetes Mellitus
Acronym: SDM
Status: Completed | Type: Observational
Sponsor: Evangelisches Krankenhaus Bielefeld gGmbH (Other)
Responsible Party: Barzu Cristian, Barzu Cristian
Other Study IDs: EvKB Barzu; DRKS00000470 (Other: German Clinical Trials Register)
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Stroke; Diabetes Mellitus
Keywords: Diabetes mellitus; Stroke
MeSH Terms: conditions — Stroke; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HbA1c ≤ 7: Stroke patients with mild diabetes mellitus HbA1c ≤ 7
- HbA1c ≥ 7,5: Stroke patients with severe diabetes mellitus HbA1c ≥ 7,5

SUMMARY:
It is to be investigated if a correlation exist between the development of the HbA1c value and the complication rate is following a stroke.

DETAILED DESCRIPTION:
The immediate objective of the study is to find out if a correlation between blood sugar control in diabetics and the incidence of complications after a stroke exists.

The study has a high practical importance because any consequences in the treatment of diabetes mellitus can be implemented without affecting costs.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients on the Stroke Unit with hyperglycemia with cerebral ischemia within the last 24 hours

Exclusion Criteria:

* Patients with intracerebral hemorrhage
* Pregnant patients
* Patients with sensory aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients on the Stroke Unit with hyperglycemia with cerebral ischemia within the last 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Functional outcome six months after the cerebral ischemia | six months
  Functional outcome for the National Institutes of Health Stroke scale, the Barthel Index and Modified Ranking Scala six months after the cerebral ischemia.

SECONDARY OUTCOMES:
Additional cerebral ischemia | six months
  Additional cerebral ischemia six months after the first cerebral ischemia
Mortality | sixt months
  Mortality in the first 6 months after the primary cerebral ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Barzu, MD, Principal Investigator — Evangelisches Krankenhaus Bielefeld, Germany
Locations (1):
- Evangelisches Krankenhaus, Bielefeld, Germany